CLINICAL TRIAL: NCT06642532
Title: A Prospective Observational Study of Transcranial Doppler Ultrasound in the Assessment of Cerebral Blood Flow After Polyetheretherketone Cranioplasty
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Junfeng Feng, Chief Director of Brain Injury Center, RenJi Hospital
Other Study IDs: LY2024-093-B
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Cranial Defect; TCD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: TCD group — Transcranial Doppler ultrasound to examine bilateral hemodynamic parameters of middle cerebral artery(MCA), terminal internal carotid artery(TICA), (anterior communicating artery)ACA, and posterior cerebral artery(PCA) (Vs, Vd, Vm, PI index, RI index) from temporal window

SUMMARY:
Polyetheretherketone has become one of the most important material choices for cranioplasty surgery. It has been shown that conventional ultrasound can be performed through the polyetheretherketone material for the examination of brain tissue and ventricular morphology. Transcranial doppler ultrasound can obtain good images of cerebral hemodynamic parameters in patients through polyetheretherketone-covered temporal window. This trial is a clinical prospective observational study in which cases treated with polyetheretherketone cranioplasty, and transcranial doppler ultrasonography is performed preoperatively and 10 days postoperatively, and data were collected mainly including bilateral hemodynamic parameters of middle cerebral artery(MCA), terminal internal carotid artery(TICA), (anterior communicating artery)ACA, and posterior cerebral artery(PCA) (Vs, Vd, Vm, PI index, RI index) from temporal window.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older;
2. Proposed polyetheretherketone cranioplasty;
3. Incomplete cranial bone in the lateral temporal window;
4. Signed informed consent for surgery and informed consent for research.

Exclusion Criteria:

1)Although cranioplasty is proposed, the cranial bone in the temporal region is intact.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age of 18 years or older;
  2. Proposed polyetheretherketone cranioplasty;
  3. Incomplete cranial bone in the lateral temporal window.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
transcranial doppler ultrasonography parameters before and after cranioplasty | 6 months
  transcranial doppler ultrasonography's hemodynamic parameters: Pulse Index（PI） of middle cerebral artery(MCA), terminal internal carotid artery(TICA), anterior communicating artery(ACA), and posterior cerebral artery(PCA) from bilateral temporal window before and after polyetheretherketone cranioplasty. PI=（Vs - Vd ）/ Vm。

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Neurosurgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Department of Neurosurgery, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No